CLINICAL TRIAL: NCT02474082
Title: A Randomized, Controlled, Multicenter, Open-label Study With Blinded Assessment of the Efficacy of Subcutaneous Secukinumab Compared to Fumaderm® in Adults With Moderate to Severe Plaque Psoriasis.
Brief Title: Study of Secukinumab Compared to Fumaderm® in Adults With Moderate to Severe Psoriasis.
Acronym: PRIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAIN457ADE06
Record Dates: First submitted 2015-04-16; First posted 2015-06-17 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab; fumaric acid; Fumarates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secukinumab (Experimental): Patients in treatment arm A will receive a dose of 300 mg secukinumab administered as 2 subcutaneous injections of 150 mg in a SensoReady pen (i.e. 2 x 150 mg) at weeks 0, 1, 2, 3, 4, 8, 12, 16 and 20.
  Interventions: Biological: Secukinumab
- Fumaric acid (initial and maintenance therapy) (Active Comparator): Participants were daily self-administered with fumaric acid derivatives initial and maintenance therapy in dosetitrated scheme as per protocol. Dose was up-titrated weekly (1 tablet/day) until objective was achieved or until tapering was required or until the maximum dose of 2 tablets each at morning, noon and evening was reached, whichever occurred earlier.
  Interventions: Drug: Fumaric acid

INTERVENTIONS:
Biological: Secukinumab — Secukinumab 150 mg, 1 ml liquid formulation in a pre-filled pen for s.c. injection
  Other Names: AIN457
  Arms: Secukinumab
Drug: Fumaric acid — Fumaric acid initial therapy (tablet contains 30 mg dimethylfumarate, 67 mg ethylhydrogenfumarate calcium salt, 5 mg ethylhydrogenfumarate magnesium salt, 3 mg ethylhydrogenfumarate zinc salt) and Fumaric acid maintenance therapy (tablet contains 120 mg dimethylfumarate, 87 mg ethylhydrogenfumarate calcium salt, 5 mg ethylhydrogenfumarate magnesium salt, 3 mg ethylhydrogenfumarate zinc salt)
  Other Names: Fumarate, Fumaric acid, Fumaric acid esters
  Arms: Fumaric acid (initial and maintenance therapy)

SUMMARY:
This is a randomized, controlled, multicenter, open-label study with blinded assessment of the efficacy of subcutaneous secukinumab compared to Fumaderm®, in 200 adults with moderate to severe plaque type psoriasis who are candidates for systemic therapy. The study consists of 2 periods: a screening period of at least one week and up to four weeks, and a treatment period of 24 weeks. During the screening period eligibility of the patients is confirmed. Eligible patients are randomized 1:1 to treatment arm A or B at week 0. Patients in treatment arm A receive secukinumab administered at weeks 0, 1, 2, 3, 4, 8, 12, 16 and 20 and are followed up for assessments of the study endpoints until week 24. Patients in treatment arm B receive daily doses of Fumaderm® p.o.. Safety and efficacy measurements of secukinumab and Fumaderm® will be performed throughout the study and up to week 24.

ELIGIBILITY:
Inclusion Criteria:

* Men or women must be at least 18 years of age at the time of screening
* Chronic plaque-type psoriasis diagnosed for at least 6 months before randomization Patients with moderate to severe plaque psoriasis who are candidates for systemic therapy as defined at randomization by:
* PASI score of >10
* Affected body surface area (BSA) > 10%
* DLQI >10
* Inadequate response, intolerance or contraindication to topical psoriasis treatment as documented in the patient's medical history or reported by the patient or determined by the investigator at screening.

Exclusion Criteria (abbreviated):

* Previous systemic treatment of plaque psoriasis or known contraindication for systemic therapy at baseline
* Ongoing use of other prohibited psoriasis and non-psoriasis treatment.
* Clinically important active infections or infestations, chronic, recurrent or latent infections or infestations
* Patients with severe liver diseases
* Patients with severe gastrointestinal diseases including but not limited to ventricular and duodenal ulcers
* Patients with severe kidney diseases or serum creatinine above 1 x ULN
* Patients with known hematological disease or lab abnormalities
* Pregnancy, breast feeding, or unwillingness/inability to use appropriate measures of contraception (if necessary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- Germany (25):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Quedlinburg
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Selters
  - Novartis Investigative Site, Stade

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 202 (secukinumab: 105 and fumaric acid derivatives: 97) participants were randomized in the study out of which 200 (secukinumab: 105 and fumaric acid derivatives: 95) received treatment. 2 participants were discontinued from the study due to non-compliance with study treatment (1) and withdrawal of informed consent (1).
Groups:
- Secukinumab: Participants were self-administered subcutaneously (s.c.) with a dose of 300 milligrams (mg) of secukinumab at weeks 0, 1, 2, 3, 4, 8, 12, 16 and 20. Secukinumab was injected in non-affected areas of the skin at front of thighs or lower abdomen (but not the area 5 centimeters (cm) around the navel).
- Fumaric Acid (Initial and Maintenance Therapy): Participants were daily self-administered with fumaric acid derivatives initial and maintenance therapy in dose-titrated scheme as per protocol. Dose was up-titrated weekly (1 tablet/day) until objective was achieved or until tapering was required or until the maximum dose of 2 tablets each at morning, noon and evening was reached, whichever occurred earlier.
Period: Overall Study
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Started | 105 | 97
Full Analysis Set (FAS) | 105 | 95
Completed | 99 | 43
Not Completed | 6 | 54
Not completed — Adverse Event | 2 | 32
Not completed — Withdrawal of informed consent | 1 | 11
Not completed — Lost to Follow-up | 2 | 2
Not completed — Dose tapering not achieved | 0 | 4
Not completed — Participant/guardian decision | 1 | 2
Not completed — Non-compliance with study treatment | 0 | 2
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Secukinumab: Participants were self-administered s.c. with a dose of 300 mg of secukinumab at weeks 0, 1, 2, 3, 4, 8, 12, 16 and 20. Secukinumab was injected in non-affected areas of the skin at front of thighs or lower abdomen (but not the area 5 cm around the navel).
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy) | Total
Number analyzed (Participants) | 105 | 97 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 90 | 188
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (14.2) | 42.4 (13.2) | 42.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 65 | 60 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 75 Response at Week 24
Description: PASI score is an average degree of severity of signs in head [H], trunk [T], upper limbs [U] and lower limbs [L], assessed separately for erythema [E], thickening (plaque elevation, induration) [I], and scaling (desquamation) [D]. Area [A] covered by lesions on each body region was estimated as a percentage (%) of total area of that particular body region and was assigned a score of 0=0%; 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100%. The head and neck, upper limbs, trunk and lower limbs correspond to approximately 10%, 20%, 30% and 40% of the body surface area, respectively. PASI score was calculated as: PASI = 0.1(EH+IH+DH) AH + 0.2(EU+IU+DU) AU + 0.3(ET+IT+DT) AT + 0.4(EL+IL+DL) AL. PASI scores can range from 0 (no signs) to a maximum of 72.0. PASI 75 responders were participants who achieved >=75% improvement (reduction) in PASI score compared to baseline.
Time Frame: Baseline, Week 24
Population: The analysis was performed in Full analysis set (FAS) population, defined as all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants | 89.52 | 33.68
Statistical Analysis 1: Comparison: Secukinumab vs Fumaric Acid (Initial and Maintenance Therapy); Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 16.61, 95% CI 2-sided [7.79 to 35.40]

2. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 50 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: PASI score is an average degree of severity of signs in head [H], trunk [T], upper limbs [U] and lower limbs [L], assessed separately for erythema [E], thickening (plaque elevation, induration) [I], and scaling (desquamation) [D]. Area [A] covered by lesions on each body region was estimated as a percentage (%) of total area of that particular body region and was assigned a score of 0=0%; 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100%. The head and neck, upper limbs, trunk and lower limbs correspond to approximately 10%, 20%, 30% and 40% of the body surface area, respectively. PASI score was calculated as: PASI = 0.1(EH+IH+DH) AH + 0.2(EU+IU+DU) AU + 0.3(ET+IT+DT) AT + 0.4(EL+IL+DL) AL. PASI scores can range from 0 (no signs) to a maximum of 72.0. PASI 50 responders were participants who achieved >=50% improvement (reduction) in PASI score compared to baseline.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed in FAS population. Here 'number analyzed' signifies participants evaluable for PASI 50 at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 105 | 91
  Week 1 | 9.5 | 1.1
  Week 2 | 37.1 | 6.3
  Week 3 | 63.8 | 10.5
  Week 4 | 81.9 | 14.7
  Week 6 | 93.3 | 28.4
  Week 8) | 96.2 | 41.1
  Week 12 | 97.1 | 56.8
  Week 16 | 98.1 | 60.0
  Week 20 | 98.1 | 61.1
  Week 24 | 98.1 | 61.1

3. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 75 Response at Week 1, 2, 3, 4, 6, 8, 12, 16 and 20
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16 and 20
Population: The analysis was performed in FAS population. Here 'number analyzed' signifies participants evaluable for PASI 75 at week 1, 2, 3, 4, 6, 8, 12, 16 and 20.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 105 | 91
  Week 1 | 0 | 0
  Week 2 | 5.7 | 0
  Week 3 | 24.8 | 0
  Week 4 | 47.6 | 1.1
  Week 6 | 69.5 | 2.1
  Week 8 | 80.0 | 8.4
  Week 12 | 87.6 | 21.1
  Week 16 | 88.6 | 27.4
  Week 20 | 88.6 | 36.8

4. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 90 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: PASI score is an average degree of severity of signs in head [H], trunk [T], upper limbs [U] and lower limbs [L], assessed separately for erythema [E], thickening (plaque elevation, induration) [I], and scaling (desquamation) [D]. Area [A] covered by lesions on each body region was estimated as a percentage (%) of total area of that particular body region and was assigned a score of 0=0%; 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100%. The head and neck, upper limbs, trunk and lower limbs correspond to approximately 10%, 20%, 30% and 40% of the body surface area, respectively. PASI score was calculated as: PASI = 0.1(EH+IH+DH) AH + 0.2(EU+IU+DU) AU + 0.3(ET+IT+DT) AT + 0.4(EL+IL+DL) AL. PASI scores can range from 0 (no signs) to a maximum of 72.0. PASI 90 responders were participants who achieved >=90% improvement (reduction) in PASI score compared to baseline.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed in FAS population. Here 'number analyzed' signifies participants evaluable for PASI 90 at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 105 | 91
  Week 1 | 0 | 0
  Week 2 | 1.9 | 0
  Week 3 | 2.9 | 0
  Week 4 | 17.1 | 0
  Week 6 | 32.4 | 0
  Week 8 | 46.7 | 1.1
  Week 12 | 63.8 | 2.1
  Week 16 | 68.6 | 8.4
  Week 20 | 75.2 | 14.7
  Week 24 | 75.2 | 18.9

5. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 100 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: PASI score is an average degree of severity of signs in head [H], trunk [T], upper limbs [U] and lower limbs [L], assessed separately for erythema [E], thickening (plaque elevation, induration) [I], and scaling (desquamation) [D]. Area [A] covered by lesions on each body region was estimated as a percentage (%) of total area of that particular body region and was assigned a score of 0=0%; 1=1-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100%. The head and neck, upper limbs, trunk and lower limbs correspond to approximately 10%, 20%, 30% and 40% of the body surface area, respectively. PASI score was calculated as: PASI = 0.1(EH+IH+DH) AH + 0.2(EU+IU+DU) AU + 0.3(ET+IT+DT) AT + 0.4(EL+IL+DL) AL. PASI scores can range from 0 (no signs) to a maximum of 72.0. PASI 100 responders were participants who achieved complete clearance of psoriasis (PASI=0).
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed in FAS population. Here 'number analyzed' signifies participants evaluable for PASI 100 at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 105 | 91
  Week 1 | 0 | 0
  Week 2 | 0 | 0
  Week 3 | 0 | 0
  Week 4 | 3.8 | 0
  Week 6 | 7.6 | 0
  Week 8 | 15.2 | 0
  Week 12 | 28.6 | 0
  Week 16 | 37.1 | 0
  Week 20 | 41.0 | 0
  Week 24 | 43.8 | 3.2

6. Secondary Outcome: Body Surface Area (BSA) at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: The Body surface area (BSA) affected by plaque-type psoriasis was the total of percentages of areas affected, including head, trunk, upper limbs and lower limbs. Each reported percentage was multiplied by its respective body region corresponding factor (head = 0.1, trunk = 0.3, upper limbs = 0.2, lower limbs = 0.4). The resulting four percentages were added to estimate the total BSA affected by plaque-type psoriasis.
Time Frame: Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed in FAS population. Here 'number analyzed' signifies participants evaluable for BSA at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Mean (Standard Deviation); unit: Percentage of area
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of area
  Week 1: number analyzed (Participants) | 105 | 94
  Week 1 | 23.8 (12.82) | 23.2 (14.11)
  Week 2: number analyzed (Participants) | 105 | 91
  Week 2 | 20.1 (12.25) | 22.5 (14.37)
  Week 3: number analyzed (Participants) | 105 | 89
  Week 3 | 17.0 (11.95) | 22.1 (14.33)
  Week 4: number analyzed (Participants) | 103 | 84
  Week 4 | 13.0 (11.93) | 21.6 (14.12)
  Week 6: number analyzed (Participants) | 98 | 82
  Week 6 | 9.8 (11.12) | 19.7 (13.52)
  Week 8: number analyzed (Participants) | 102 | 75
  Week 8 | 7.6 (10.19) | 17.8 (12.65)
  Week 12: number analyzed (Participants) | 103 | 67
  Week 12 | 5.2 (9.12) | 13.7 (11.60)
  Week 16: number analyzed (Participants) | 99 | 59
  Week 16 | 3.7 (6.72) | 11.4 (11.52)
  Week 20: number analyzed (Participants) | 99 | 50
  Week 20 | 2.6 (5.77) | 9.2 (11.87)
  Week 24: number analyzed (Participants) | 99 | 48
  Week 24 | 2.9 (6.43) | 7.9 (9.92)

7. Secondary Outcome: Percentage of Participants Achieving Nail Psoriasis Severity Index (NAPSI) 50 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: NAPSI was used to assess psoriatic nail involvement in participants with nail psoriasis. NAPSI score was calculated as total of nail matrix and nail bed score, ranging from 0-8 per nail. Total NAPSI score ranges from 0 to 80 for all fingernails. Each nail was divided with imaginary horizontal and longitudinal lines into quadrants. Each nail was given a score of 0 - 4 for nail matrix and nail bed psoriasis 0-4 (0: for none, 1: for 1 quadrant, 2: for 2 quadrants, 3: for 3 quadrants, 4: for all 4 quadrants), based on presence of any feature of nail psoriasis in that quadrant. Nail matrix psoriasis feature includes: pitting, leukonychia red spots in lunula, crumbling. Nail bed psoriasis feature includes: onycholysis, splinter hemorrhages, subungual hyperkeratosis, "oil drop" (salmon patch dyschroma). NPASI 50 responders were participants who achieved >=50% improvement (reduction) in NPASI score compared to baseline.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population. Here 'number analyzed' signifies participants evaluable for NAPSI 50 at week 1, 2, 3, 4, 5, 6, 7,12,16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 49
  Week 1 | 1.8 | 4.1
  Week 2: number analyzed (Participants) | 56 | 49
  Week 2 | 3.6 | 8.2
  Week 3: number analyzed (Participants) | 56 | 49
  Week 3 | 5.4 | 10.2
  Week 4: number analyzed (Participants) | 56 | 49
  Week 4 | 7.1 | 12.2
  Week 6: number analyzed (Participants) | 56 | 49
  Week 6 | 19.6 | 10.2
  Week 8: number analyzed (Participants) | 56 | 49
  Week 8 | 23.2 | 8.2
  Week 12: number analyzed (Participants) | 56 | 49
  Week 12 | 41.1 | 12.2
  Week 16: number analyzed (Participants) | 56 | 49
  Week 16 | 51.8 | 10.2
  Week 20: number analyzed (Participants) | 56 | 49
  Week 20 | 62.5 | 18.4
  Week 24: number analyzed (Participants) | 56 | 49
  Week 24 | 67.9 | 18.4

8. Secondary Outcome: Percentage of Participants Achieving Nail Psoriasis Severity Index (NAPSI) 75 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: NAPSI was used to assess psoriatic nail involvement in participants with nail psoriasis. NAPSI score was calculated as total of nail matrix and nail bed score, ranging from 0-8 per nail. Total NAPSI score ranges from 0 to 80 for all fingernails. Each nail was divided with imaginary horizontal and longitudinal lines into quadrants. Each nail was given a score of 0 - 4 for nail matrix and nail bed psoriasis 0-4 (0: for none, 1: for 1 quadrant, 2: for 2 quadrants, 3: for 3 quadrants, 4: for all 4 quadrants), based on presence of any feature of nail psoriasis in that quadrant. Nail matrix psoriasis feature includes: pitting, leukonychia red spots in lunula, crumbling. Nail bed psoriasis feature includes: onycholysis, splinter hemorrhages, subungual hyperkeratosis, "oil drop" (salmon patch dyschroma). NPASI 75 responders were participants who achieved >=75% improvement (reduction) in NPASI score compared to baseline.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population. Here 'number analyzed' signifies participants evaluable for NAPSI 75 at week 1, 2, 3, 4, 5, 6, 8,12,16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 49
  Week 1 | 1.8 | 0
  Week 2: number analyzed (Participants) | 56 | 49
  Week 2 | 1.8 | 2.0
  Week 3: number analyzed (Participants) | 56 | 49
  Week 3 | 5.4 | 2.0
  Week 4: number analyzed (Participants) | 56 | 49
  Week 4 | 7.1 | 2.0
  Week 6: number analyzed (Participants) | 56 | 49
  Week 6 | 8.9 | 2.0
  Week 8: number analyzed (Participants) | 56 | 49
  Week 8 | 17.9 | 2.0
  Week 12: number analyzed (Participants) | 56 | 49
  Week 12 | 28.6 | 2.0
  Week 16: number analyzed (Participants) | 56 | 49
  Week 16 | 30.4 | 2.0
  Week 20: number analyzed (Participants) | 56 | 49
  Week 20 | 44.6 | 6.1
  Week 24: number analyzed (Participants) | 56 | 49
  Week 24 | 53.6 | 4.1

9. Secondary Outcome: Percentage of Participants Achieving Nail Psoriasis Severity Index (NAPSI) 90 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: NAPSI was used to assess psoriatic nail involvement in participants with nail psoriasis. NAPSI score was calculated as total of nail matrix and nail bed score, ranging from 0-8 per nail. Total NAPSI score ranges from 0 to 80 for all fingernails. Each nail was divided with imaginary horizontal and longitudinal lines into quadrants. Each nail was given a score of 0 - 4 for nail matrix and nail bed psoriasis 0-4 (0: for none, 1: for 1 quadrant, 2: for 2 quadrants, 3: for 3 quadrants, 4: for all 4 quadrants), based on presence of any feature of nail psoriasis in that quadrant. Nail matrix psoriasis feature includes: pitting, leukonychia red spots in lunula, crumbling. Nail bed psoriasis feature includes: onycholysis, splinter hemorrhages, subungual hyperkeratosis, "oil drop" (salmon patch dyschroma). NPASI 90 responders were participants who achieved >=90% improvement (reduction) in NPASI score compared to baseline.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population. Here 'number analyzed' signifies the participants evaluable for NAPSI 90 response at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 49
  Week 1 | 1.8 | 0
  Week 2: number analyzed (Participants) | 56 | 49
  Week 2 | 1.8 | 0
  Week 3: number analyzed (Participants) | 56 | 49
  Week 3 | 0 | 0
  Week 4: number analyzed (Participants) | 56 | 49
  Week 4 | 3.6 | 0
  Week 6: number analyzed (Participants) | 56 | 49
  Week 6 | 3.6 | 0
  Week 8: number analyzed (Participants) | 56 | 49
  Week 8 | 7.1 | 2.0
  Week 12: number analyzed (Participants) | 56 | 49
  Week 12 | 14.3 | 2.0
  Week 16: number analyzed (Participants) | 56 | 49
  Week 16 | 21.4 | 2.0
  Week 20: number analyzed (Participants) | 56 | 49
  Week 20 | 26.8 | 4.1
  Week 24: number analyzed (Participants) | 56 | 49
  Week 24 | 35.7 | 4.1

10. Secondary Outcome: Percentage of Participants Achieving Nail Psoriasis Severity Index (NAPSI) 100 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: NAPSI was used to assess psoriatic nail involvement in participants with nail psoriasis. NAPSI score was calculated as total of nail matrix and nail bed score, ranging from 0-8 per nail. Total NAPSI score ranges from 0 to 80 for all fingernails. Each nail was divided with imaginary horizontal and longitudinal lines into quadrants. Each nail was given a score of 0 - 4 for nail matrix and nail bed psoriasis 0-4 (0: for none, 1: for 1 quadrant, 2: for 2 quadrants, 3: for 3 quadrants, 4: for all 4 quadrants), based on presence of any feature of nail psoriasis in that quadrant. Nail matrix psoriasis feature includes: pitting, leukonychia red spots in lunula, crumbling. Nail bed psoriasis feature includes: onycholysis, splinter hemorrhages, subungual hyperkeratosis, "oil drop" (salmon patch dyschroma). NPASI 100 responders were participants who PASI 100 responders were participants who achieved complete clearance of psoriasis.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population. Here 'number analyzed' signifies the participants evaluable for NAPSI 100 response at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 49
  Week 1 | 1.8 | 0
  Week 2: number analyzed (Participants) | 56 | 49
  Week 2 | 0 | 0
  Week 3: number analyzed (Participants) | 56 | 49
  Week 3 | 0 | 0
  Week 4: number analyzed (Participants) | 56 | 49
  Week 4 | 3.6 | 0
  Week 6: number analyzed (Participants) | 56 | 49
  Week 6 | 3.6 | 0
  Week 8: number analyzed (Participants) | 56 | 49
  Week 8 | 5.4 | 2.0
  Week 12: number analyzed (Participants) | 56 | 49
  Week 12 | 10.7 | 2.0
  Week 16: number analyzed (Participants) | 56 | 49
  Week 16 | 19.6 | 2.0
  Week 20: number analyzed (Participants) | 56 | 49
  Week 20 | 19.6 | 2.0
  Week 24: number analyzed (Participants) | 56 | 49
  Week 24 | 23.2 | 2.0

11. Secondary Outcome: Number of Participants With Investigator's Global Assessment (IGA Mod 2011) at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: IGA mod 2011 is a global static severity rating scale referring exclusively to the participant's disease state at the time of the assessments and don't attempt comparison with participant's any previous disease states at baseline or visit. IGA mod 2011 has a scale of 0-4 with the lower scores correlating to better performance. Scores used were: 0/Clear: no signs of psoriasis, Post-inflammatory hyperpigmentation may be present; 1/almost clear: Normal to pink coloration of lesions/no thickening/no to minimal focal scaling; 2/Mild: Pink to light red coloration/just detectable to mild thickening/predominantly fine scaling; 3/Moderate: Dull bright red, clearly distinguishable erythema/clearly distinguishable to moderate thickening/moderate scaling; 4/Severe: Bright to deep dark red coloration/severe thickening with hard edges/severe or coarse scaling covering almost all or all lesions.
Time Frame: Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed in FAS population. Here 'number analyzed' signifies the participants evaluable for IGA mod 2011 at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Participants
  Week 1: Clear: number analyzed (Participants) | 105 | 94
  Week 1: Clear | 0 | 0
  Week 1: Almost Clear: number analyzed (Participants) | 105 | 94
  Week 1: Almost Clear | 0 | 0
  Week 1: Mild: number analyzed (Participants) | 105 | 94
  Week 1: Mild | 18 | 8
  Week 1: Moderate: number analyzed (Participants) | 105 | 94
  Week 1: Moderate | 65 | 58
  Week 1: Severe: number analyzed (Participants) | 105 | 94
  Week 1: Severe | 22 | 28
  Week 2: Clear: number analyzed (Participants) | 105 | 91
  Week 2: Clear | 0 | 0
  Week 2: Almost Clear: number analyzed (Participants) | 105 | 91
  Week 2: Almost Clear | 6 | 0
  Week 2: Mild: number analyzed (Participants) | 105 | 91
  Week 2: Mild | 38 | 15
  Week 2: Moderate: number analyzed (Participants) | 105 | 91
  Week 2: Moderate | 49 | 56
  Week 2: Severe: number analyzed (Participants) | 105 | 91
  Week 2: Severe | 12 | 20
  Week 3: Clear: number analyzed (Participants) | 105 | 89
  Week 3: Clear | 0 | 0
  Week 3: Almost Clear: number analyzed (Participants) | 105 | 89
  Week 3: Almost Clear | 14 | 1
  Week 3: Mild: number analyzed (Participants) | 105 | 89
  Week 3: Mild | 51 | 18
  Week 3: Moderate: number analyzed (Participants) | 105 | 89
  Week 3: Moderate | 35 | 51
  Week 3: Severe: number analyzed (Participants) | 105 | 89
  Week 3: Severe | 5 | 19
  Week 4: Clear: number analyzed (Participants) | 103 | 84
  Week 4: Clear | 4 | 0
  Week 4: Almost Clear: number analyzed (Participants) | 103 | 84
  Week 4: Almost Clear | 31 | 1
  Week 4: Mild: number analyzed (Participants) | 103 | 84
  Week 4: Mild | 46 | 21
  Week 4: Moderate: number analyzed (Participants) | 103 | 84
  Week 4: Moderate | 19 | 46
  Week 4: Severe: number analyzed (Participants) | 103 | 84
  Week 4: Severe | 3 | 16
  Week 6: Clear: number analyzed (Participants) | 98 | 82
  Week 6: Clear | 9 | 0
  Week 6: Almost Clear: number analyzed (Participants) | 98 | 82
  Week 6: Almost Clear | 42 | 2
  Week 6: Mild: number analyzed (Participants) | 98 | 82
  Week 6: Mild | 39 | 26
  Week 6: Moderate: number analyzed (Participants) | 98 | 82
  Week 6: Moderate | 7 | 44
  Week 6: Severe: number analyzed (Participants) | 98 | 82
  Week 6: Severe | 1 | 10
  Week 8: Clear: number analyzed (Participants) | 102 | 75
  Week 8: Clear | 17 | 0
  Week 8: Almost Clear: number analyzed (Participants) | 102 | 75
  Week 8: Almost Clear | 52 | 4
  Week 8: Mild: number analyzed (Participants) | 102 | 95
  Week 8: Mild | 29 | 32
  Week 8: Moderate: number analyzed (Participants) | 102 | 75
  Week 8: Moderate | 2 | 34
  Week 8: Severe: number analyzed (Participants) | 102 | 75
  Week 8: Severe | 2 | 5
  Week 12: Clear: number analyzed (Participants) | 103 | 67
  Week 12: Clear | 31 | 0
  Week 12: Almost Clear: number analyzed (Participants) | 103 | 67
  Week 12: Almost Clear | 49 | 11
  Week 12: Mild: number analyzed (Participants) | 103 | 67
  Week 12: Mild | 19 | 35
  Week 12: Moderate: number analyzed (Participants) | 103 | 67
  Week 12: Moderate | 4 | 19
  Week 12: Severe: number analyzed (Participants) | 103 | 67
  Week 12: Severe | 0 | 2
  Week 16: Clear: number analyzed (Participants) | 99 | 59
  Week 16: Clear | 38 | 0
  Week 16: Almost Clear: number analyzed (Participants) | 99 | 59
  Week 16: Almost Clear | 42 | 12
  Week 16: Mild: number analyzed (Participants) | 99 | 59
  Week 16: Mild | 15 | 35
  Week 16: Moderate: number analyzed (Participants) | 99 | 59
  Week 16: Moderate | 4 | 11
  Week 16: Severe: number analyzed (Participants) | 99 | 59
  Week 16: Severe | 0 | 1
  Week 20: Clear: number analyzed (Participants) | 99 | 50
  Week 20: Clear | 43 | 0
  Week 20: Almost Clear: number analyzed (Participants) | 99 | 50
  Week 20: Almost Clear | 36 | 17
  Week 20: Mild: number analyzed (Participants) | 99 | 50
  Week 20: Mild | 18 | 24
  Week 20: Moderate: number analyzed (Participants) | 99 | 50
  Week 20: Moderate | 2 | 8
  Week 20: Severe: number analyzed (Participants) | 99 | 50
  Week 20: Severe | 0 | 1
  Week 24: Clear: number analyzed (Participants) | 99 | 48
  Week 24: Clear | 45 | 4
  Week 24: Almost Clear: number analyzed (Participants) | 99 | 48
  Week 24: Almost Clear | 36 | 21
  Week 24: Mild: number analyzed (Participants) | 99 | 48
  Week 24: Mild | 13 | 15
  Week 24: Moderate: number analyzed (Participants) | 99 | 48
  Week 24: Moderate | 5 | 7
  Week 24: Severe: number analyzed (Participants) | 99 | 48
  Week 24: Severe | 0 | 1

12. Secondary Outcome: Percentage of Participants With IGA Mod. 2011 0/1-response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: The IGA mod 2011 scale has been developed based on a previous version of the scale used in secukinumab phase II studies in collaboration with health authorities, in particular the FDA. The explanations/descriptions of the points on the scale have been improved to ensure appropriate differentiation between the points. The IGA mod 2011 used in this study is static, i.e. it refers exclusively to the subject's disease state at the time of the assessments, and does not attempt a comparison with any of the subject's previous disease states, whether at baseline or at a previous visit.IGA mod 2011 has a scale of 0-4 with the lower scores correlating to better performance. A score of 0= clear skin, 1= almost clear skin, 2=mild, 3=moderate,4=severe. IGA 0/1 responders: who achieved score of 0/1 and improved by at least 2 points on the IGA scale compared to baseline.
Time Frame: Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1 | 0 | 0
  Week 2 | 5.7 | 0
  Week 3 | 13.3 | 1.1
  Week 4 | 34.3 | 1.1
  Week 6 | 50.5 | 2.1
  Week 8 | 66.7 | 4.2
  Week 12 | 77.1 | 12.6
  Week 16 | 80.0 | 14.7
  Week 20 | 79.0 | 20.0
  Week 24 | 81.0 | 28.4

13. Secondary Outcome: Dermatology Life Quality Index (DLQI) at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life in adult subjects with skin diseases such as eczema, psoriasis, acne, and viral. The measure was self-administered and included domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. Each item had four response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" was also a valid response and was scored as 0. The DLQI total score was a sum of the 10 questions. Scores ranged from 0 to 30, with higher scores indicating greater impairment in health related quality of life.
Time Frame: Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population. Here 'number analyzed' signifies the participants evaluable for DLQI at week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Score on a scale
  Week 1: number analyzed (Participants) | 105 | 94
  Week 1 | 13.9 (5.86) | 16.3 (6.44)
  Week 2: number analyzed (Participants) | 105 | 91
  Week 2 | 10.5 (6.22) | 15.3 (6.99)
  Week 3: number analyzed (Participants) | 105 | 89
  Week 3 | 8.4 (5.96) | 14.6 (7.01)
  Week 4: number analyzed (Participants) | 102 | 84
  Week 4 | 6.6 (5.13) | 13.8 (7.23)
  Week 6: number analyzed (Participants) | 98 | 82
  Week 6 | 5.3 (5.79) | 12.4 (7.24)
  Week 8: number analyzed (Participants) | 102 | 77
  Week 8 | 4.2 (4.75) | 11.0 (7.16)
  Week 12: number analyzed (Participants) | 103 | 67
  Week 12 | 3.1 (4.41) | 8.8 (7.10)
  Week 16: number analyzed (Participants) | 99 | 59
  Week 16 | 2.7 (3.95) | 6.8 (6.05)
  Week 20: number analyzed (Participants) | 98 | 50
  Week 20 | 2.5 (3.84) | 5.9 (5.67)
  Week 24: number analyzed (Participants) | 99 | 48
  Week 24 | 2.0 (3.58) | 5.4 (5.56)

14. Secondary Outcome: Percentage of Participants With DLQI 0/1 Response at Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Description: DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life in adult subjects with skin diseases such as eczema, psoriasis, acne, and viral. The measure was self-administered and included domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. Each item had four response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" was also a valid response and was scored as 0. The DLQI total score was a sum of the 10 questions. Scores ranged from 0 to 30, with higher scores indicating greater impairment in health related quality of life. DLQI 0/1 response was the achievement of a DLQI score of 0 or 1.
Time Frame: Week 1, 2, 3, 4, 6, 8, 12, 16, 20 and 24
Population: The analysis was performed on FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Week 1 | 0 | 0
  Week 2 | 3.8 | 1.1
  Week 3 | 7.6 | 0
  Week 4 | 19.0 | 2.1
  Week 6 | 30.5 | 4.2
  Week 8 | 40.0 | 6.3
  Week 12 | 57.1 | 10.5
  Week 16 | 59.0 | 14.7
  Week 20 | 64.8 | 15.8
  Week 24 | 71.4 | 25.3

15. Secondary Outcome: Percentage of Participants With Short Form 36 (SF-36) Response at Week 4, 16 and 24
Description: SF-36 is a generic indicator of health status for use in population surveys and evaluative studies of health policy. The SF-36 included 36 items in a Likert-type or forced-choice format measured on eight dimensions. The scores for each domain range from 0 to 100, with high scores indicating a better status. SF-36 responder is defined as subject reaching at least an improvement of minimum important difference (MID). The SF-36 measure dimensions and their MID includes:
  * Physical Functioning:4.3
  * Role-Physical: 3.4
  * Bodily Pain: 6.2
  * General Health: 7.2
  * Vitality: 6.2
  * Social Functioning: 6.9
  * Role-Emotional: 4.5
  * Mental Health: 6.2
  Two component scores and their MID which were derived from the above mentioned 8 domains includes-:
  * Physical component summary: 3.4
  * Mental component summary: 4.6
Time Frame: Week 4, 16 and 24
Population: The analysis was performed on FAS population. Here 'number analyzed' signifies the participants evaluable for SF-36 response at week 4, 16 and 24
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Number analyzed (Participants) | 105 | 95
Percentage of participants
  Physical Component Summary Week 4: number analyzed (Participants) | 97 | 88
  Physical Component Summary Week 4 | 38.1 | 26.1
  Mental component summary Week 4: number analyzed (Participants) | 97 | 88
  Mental component summary Week 4 | 41.2 | 36.4
  Physical functioning scale Week 4: number analyzed (Participants) | 102 | 92
  Physical functioning scale Week 4 | 24.5 | 19.6
  Role physical scale Week 4: number analyzed (Participants) | 104 | 93
  Role physical scale Week 4 | 44.2 | 23.7
  Bodily pain scale Week 4 | 53.3 | 31.6
  General health scale Week 4: number analyzed (Participants) | 102 | 95
  General health scale Week 4 | 32.4 | 21.1
  Vitality scale Week 4: number analyzed (Participants) | 104 | 93
  Vitality scale Week 4 | 31.7 | 20.4
  Social functioning scale Week 4: number analyzed (Participants) | 102 | 94
  Social functioning scale Week 4 | 39.2 | 27.7
  Role emotional scale Week 4: number analyzed (Participants) | 104 | 95
  Role emotional scale Week 4 | 41.3 | 34.7
  Mental health scale Week 4 | 33.3 | 32.6
  Physical Component Summary Week 16: number analyzed (Participants) | 97 | 88
  Physical Component Summary Week 16 | 52.6 | 39.8
  Mental component summary Week 16: number analyzed (Participants) | 97 | 88
  Mental component summary Week 16 | 63.9 | 46.6
  Physical functioning scale Week 16: number analyzed (Participants) | 102 | 92
  Physical functioning scale Week 16 | 36.3 | 31.5
  Role physical scale Week 16: number analyzed (Participants) | 104 | 93
  Role physical scale Week 16 | 52.9 | 36.6
  Bodily pain scale Week 16 | 63.8 | 45.3
  General health scale Week 16: number analyzed (Participants) | 102 | 95
  General health scale Week 16 | 38.2 | 22.1
  Vitality scale Week 16: number analyzed (Participants) | 104 | 93
  Vitality scale Week 16 | 45.2 | 23.7
  Social functioning scale Week 16: number analyzed (Participants) | 102 | 94
  Social functioning scale Week 16 | 57.8 | 41.5
  Role emotional scale Week 16: number analyzed (Participants) | 104 | 95
  Role emotional scale Week 16 | 56.7 | 43.2
  Mental health scale Week 16 | 54.3 | 42.1
  Physical Component Summary Week 24: number analyzed (Participants) | 97 | 88
  Physical Component Summary Week 24 | 57.7 | 43.2
  Mental component summary Week 24: number analyzed (Participants) | 97 | 88
  Mental component summary Week 24 | 63.9 | 50.0
  Physical functioning scale Week 24: number analyzed (Participants) | 102 | 92
  Physical functioning scale Week 24 | 38.2 | 31.5
  Role physical scale Week 24: number analyzed (Participants) | 104 | 93
  Role physical scale Week 24 | 52.9 | 37.6
  Bodily pain scale Week 24 | 64.8 | 49.5
  General health scale Week 24: number analyzed (Participants) | 102 | 95
  General health scale Week 24 | 41.2 | 21.1
  Vitality scale Week 24: number analyzed (Participants) | 104 | 93
  Vitality scale Week 24 | 48.1 | 29.0
  Social functioning scale Week 24: number analyzed (Participants) | 102 | 94
  Social functioning scale Week 24 | 63.7 | 45.7
  Role emotional scale Week 24: number analyzed (Participants) | 104 | 95
  Role emotional scale Week 24 | 54.8 | 41.1
  Mental health scale Week 24 | 53.3 | 38.9

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit (up to 29 weeks).
Description: The safety analysis set consisted of all patients who took at least one dose of study treatment during the treatment period.
Arm/Group | Secukinumab | Fumaric Acid (Initial and Maintenance Therapy)
Serious Adverse Events (participants affected / at risk) | 4/105 | 4/95
Other Adverse Events (participants affected / at risk) | 75/105 | 85/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=105) | Fumaric Acid (Initial and Maintenance Therapy) (N=95)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 1 | 0
PILONIDAL CYST (Infections and infestations) | 0 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BRAIN OEDEMA (Nervous system disorders) | 1 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 2
THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=105) | Fumaric Acid (Initial and Maintenance Therapy) (N=95)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 | 17
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 5
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 5
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 | 23
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 11
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 37
DIARRHOEA (Gastrointestinal disorders) | 7 | 48
FLATULENCE (Gastrointestinal disorders) | 0 | 5
NAUSEA (Gastrointestinal disorders) | 3 | 20
VOMITING (Gastrointestinal disorders) | 2 | 7
FATIGUE (General disorders) | 4 | 6
NASOPHARYNGITIS (Infections and infestations) | 54 | 40
URINARY TRACT INFECTION (Infections and infestations) | 6 | 3
BLOOD CREATININE INCREASED (Investigations) | 1 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 4
HEADACHE (Nervous system disorders) | 15 | 15
HAEMATURIA (Renal and urinary disorders) | 6 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 7 | 8
FLUSHING (Vascular disorders) | 1 | 34
HOT FLUSH (Vascular disorders) | 1 | 7
HYPERTENSION (Vascular disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.